CLINICAL TRIAL: NCT06643520
Title: Sample Adequacy and Diagnostic Accuracy of a 22 Gauge FNB Needle vs a 19G FNB Needle for EUS-guided Liver Biopsy: a Prospective Trial
Brief Title: 19G FNB Needle vs 22G FNB Needle for EUS-Guided Liver Biopsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duzce University (Other)
Responsible Party: Principal Investigator, Salih Tokmak, Assoc.Prof. of GI, Duzce University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: EUS-LB
Record Dates: First submitted 2024-10-10; First posted 2024-10-16 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Endoscopic Ultrasonography; Liver Biopsy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 19-gauge FNB needle (Active Comparator): Biopsy samples obtained by a 19-gauge FNB needles for EUS-LB
  Interventions: Device: 19-gauge
- 22-gauge FNB needle (Experimental): Biopsy samples obtained by a 22-gauge FNB needles for EUS-LB
  Interventions: Device: 22-gauge

INTERVENTIONS:
Device: 19-gauge — All procedures will be performed under monitored endoscopist- directed anesthesia. Patients will be placed in a semi-prone position and oxygen at a rate of 3 L/min will be administered routinely
  All procedures will be performed by the same endoscopist, who performed > 500 diagnostic and interventional EUS procedures annually. A standard linear echoendoscope (EG34-J10U, Pentax Medi- cal, Hoya Corp, Japan) will be used. The patients are going to be followed up until the Modified Aldrete Score > 9 after the procedure, and then they will be discharged.
  All biopsies will be performed with a standard 19 gauge FNA needle (Trident, Micro-Tech (Nanjing) Co., Ltd, Nan) with wet suction technique. Biopsy needles will be used without stylets and primed with diluted heparin (1:1 ratio) to obtain samples by wet-suction technique to prevent clot formation. All the biopsies will be performed from the left lobe of the liver as one pass and five actuations.
  Arms: 19-gauge FNB needle
Device: 22-gauge — All procedures will be performed under monitored endoscopist- directed anesthesia. Patients will be placed in a semi-prone position and oxygen at a rate of 3 L/min will be administered routinely.
  All procedures will be performed by the same endoscopist, who performed > 500 diagnostic and interventional EUS procedures annually. A standard linear echoendoscope (EG34-J10U, Pentax Medi- cal, Hoya Corp, Japan) will be used. The patients are going to be followed up until the Modified Aldrete Score > 9 after the procedure, and then they will be discharged.
  All biopsies will be performed with a standard 22 gauge FNA needle (Trident, Micro-Tech (Nanjing) Co., Ltd, Nan) with wet suction technique. Biopsy needles will be used without stylets and primed with diluted heparin (1:1 ratio) to obtain samples by wet-suction technique to prevent clot formation. All the biopsies will be performed from the left lobe of the liver as one pass and five actuations.
  Arms: 22-gauge FNB needle

SUMMARY:
EUS-guided liver biopsy (EUS-LB) is increasingly used to diagnose patients with liver disease, especially in anxious patients who need sedation. There is an ongoing debate about the optimal needle size for EUS-LB. Some clinicians prefer a thinner 22-gauge biopsy needle because they presume it to be safer, and some studies show that their performance is the same as a thicker 19-gauge needle. However, some other studies show that the adequacy and diagnostic accuracy of a 19-gauge needle is better, and the rates of adverse events are the same. In this study, we aimed to compare the adequacy and diagnostic accuracy of samples obtained by the same endoscopist from the same liver lobe during the same session.

ELIGIBILITY:
Inclusion Criteria:

* All patients with unexplained elevation of liver enzymes and suspected hepatic paranchymal disease

Exclusion Criteria:

* Patients who had malignancy
* Patients who have decompensated cirrhosis
* Presence of ascites
* Patients with coagulopathy (platelets < 50.000 μ/ mL and INR > 1.5)
* The use of anticoagulant agents
* Pregnancy
* Unable to provide written informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-03-01 (Actual); Study Completion 2025-04-01 (Actual)

PRIMARY OUTCOMES:
Sample adequacy | 1 month
  The sample must have at least 11 complete portal tracts and the length of the longest specimen should be at least 15mm

SECONDARY OUTCOMES:
Adverse events | 1 week
  The rates of adverse events will be recorded. According to the American Society of Gastrointestinal Endoscopy lexicon, an adverse event is "… an event preventing the completion of the planned procedure and/or results in admission to the hospital, prolonga- tion of existing hospital stay, another procedure (needing sedation/anesthesia), or subsequent medical consultation."

CONTACTS AND LOCATIONS:
Locations (1):
- Duzce University, Düzce, Düzce, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah RM, Schmidt J, John E, Rastegari S, Acharya P, Kedia P. Superior Specimen and Diagnostic Accuracy with Endoscopic Ultrasound-Guided Liver Biopsies Using 19-Gauge versus 22-Gauge Core Needles. Clin Endosc. 2021 Sep;54(5):739-744. doi: 10.5946/ce.2020.212. Epub 2020 Nov 13. PMID 33189102
- [Background] Dalal A, Kamat N, Patil G, Vadgaonkar A, Parekh S, Vora S, Maydeo A. Comparison of diagnostic outcomes, safety, and cost of Franseen-tip 19G versus 22G needles for endoscopic ultrasound-guided liver biopsies. Endosc Int Open. 2024 Feb 28;12(2):E291-E296. doi: 10.1055/a-2226-1337. eCollection 2024 Feb. PMID 38420158
- [Background] Diehl DL, Sangwan V, Johal AS, Khara HS, Confer B. Comparing a 19-gauge fine-needle biopsy needle with a 22-gauge fine-needle biopsy needle for EUS-guided liver biopsy sampling: a prospective randomized study. Gastrointest Endosc. 2024 Jun;99(6):931-937. doi: 10.1016/j.gie.2023.12.022. Epub 2023 Dec 21. PMID 38141686